CLINICAL TRIAL: NCT06489080
Title: Survival and cArdiovascular eVents in Patients With Acute Myocardial Infarction in Peking UNiversity First Hospital: A lonG-term Cohort Study
Brief Title: Survival and cArdiovascular eVents in Patients With Acute Myocardial Infarction
Acronym: SAVING
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jianping LI, Director of Department of Cardiology, Peking University First Hospital
Other Study IDs: 2024yan097-002
Record Dates: First submitted 2024-06-23; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease
Keywords: Acute Myocardial Infarction; Coronary Artery Disease; cohort study
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective and prospective cohort study aims to establish a long-term follow-up cohort of patients with acute myocardial infarction, and combine multi-omics studies, wearable devices, artificial intelligence technology, etc., to describe the clinical characteristics of patients with acute myocardial infarction and the changing trend of treatment strategies, and analyze the related influencing factors. Explore new biomarkers and indicators affecting recurrent cardiovascular events for accurate risk stratification and risk prediction; To evaluate the factors affecting lifestyle intervention, drug efficacy and safety, and their impact on outcome, and improve chronic disease management mode, in order to improve the quality of life and prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction is diagnosed meets the universal definition of acute myocardial infarction

Exclusion Criteria:

* Did not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the department of Cardiology or outpatient department of Peking University First Hospital will be enrolled if they are aged ≥18 years old, meet the inclusion criteria of acute myocardial infarction and need long-term follow-up according to the judgment of doctors after informed consent. There are about 7500 retrospectively enrolled patients, and it is expected to enroll 500 patients per year.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 5 years
  Composite end points of Cardiovascular death, nonfatal myocardial infarction, nonfatal ischemic stroke

SECONDARY OUTCOMES:
Secondary Adverse Cardiovascular Events | 5 years
  All-cause death, non-cardiac death, myocardial infarction, hospitalization for coronary revascularization, hospitalization for heart failure, hospitalization for acute coronary syndrome, ischemic stroke, hemorrhagic stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Li J, Li X, Wang Q, Hu S, Wang Y, Masoudi FA, Spertus JA, Krumholz HM, Jiang L; China PEACE Collaborative Group. ST-segment elevation myocardial infarction in China from 2001 to 2011 (the China PEACE-Retrospective Acute Myocardial Infarction Study): a retrospective analysis of hospital data. Lancet. 2015 Jan 31;385(9966):441-51. doi: 10.1016/S0140-6736(14)60921-1. Epub 2014 Jun 23. PMID 24969506
- [Background] Xu H, Yang Y, Wang C, Yang J, Li W, Zhang X, Ye Y, Dong Q, Fu R, Sun H, Yan X, Gao X, Wang Y, Jia X, Sun Y, Wu Y, Zhang J, Zhao W, Sabatine MS, Wiviott SD; China Acute Myocardial Infarction Registry Investigators. Association of Hospital-Level Differences in Care With Outcomes Among Patients With Acute ST-Segment Elevation Myocardial Infarction in China. JAMA Netw Open. 2020 Oct 1;3(10):e2021677. doi: 10.1001/jamanetworkopen.2020.21677. PMID 33095249
- [Background] Hao Y, Zhao D, Liu J, Liu J, Yang N, Huo Y, Fonarow GC, Ge J, Morgan L, Ma C, Han Y, Smith SC Jr; CCC-ACS Investigators. Performance of Management Strategies With Class I Recommendations Among Patients Hospitalized With ST-Segment Elevation Myocardial Infarction in China. JAMA Cardiol. 2022 May 1;7(5):484-491. doi: 10.1001/jamacardio.2022.0117. PMID 35293976